CLINICAL TRIAL: NCT00202657
Title: Etude Observationnelle Des Valvulopathies Chez Les Patients Parkinsoniens Traites Par Pergolide Par Rapport a Une Population Temoin
Brief Title: Observational Study of Heart Valve Disease in Patients With Parkinson's Disease Treated With Pergolide
Status: Completed | Type: Observational
Sponsor: Société Française de Cardiologie (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Other Study IDs: 2005-03
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Parkinson's Disease; Pergolide
Keywords: parkinson's disease; pergolide; heart valve disease
MeSH Terms: conditions — Parkinson Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: echocardiography

SUMMARY:
The purpose of this study is to determine whether patients with Parkinson's disease and treated with pergolide have a higher risk of heart valve disease compared to patients with Parkinson's disease not treated with pergolide.

DETAILED DESCRIPTION:
Pergolide is an ergot dopamine receptor agonist with demonstrated efficacy in Parkinson's disease. Last year, two studies showed that pergolide can induce unexpected heart valve disease potentially severe and frequent. The late discovery of this unknown side effect had dramatic consequences in Parkinson's disease management and the French drug agency (AFFSAPS) has recently published guidelines for its prescription. Little is known about the prevalence and the molecular mechanisms leading to this adverse event. To determine the prevalence, evolution, and potential risk factors of pergolide-induced heart valve disease, we propose an echocardiographic observational study in parkinsonian patients taking pergolide compared to matched controls. This clinical study will be performed in the Clinical Investigation Centre in collaboration with the Institute of Cardiology of the Salpétrière Hospital

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Hoehn and Yahr score inferior or equal to 4
* treated with pergolide since more than 3 months (pergolide group)
* never treated by pergolide (control group)

Exclusion Criteria:

* Parkinson + syndrome, multiple system atrophy, supranuclear palsy
* hoehn and yahr score equal to 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Pergolide for Parkinson disease or Patients with parkinson disease not treated with Pergolide
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2005-04; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe CORVOL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Clinical Investigation Centre, Pitie-Salpetriere Hospital, Paris, France

REFERENCES:
- [Derived] Corvol JC, Anzouan-Kacou JB, Fauveau E, Bonnet AM, Lebrun-Vignes B, Girault C, Agid Y, Lechat P, Isnard R, Lacomblez L. Heart valve regurgitation, pergolide use, and parkinson disease: an observational study and meta-analysis. Arch Neurol. 2007 Dec;64(12):1721-6. doi: 10.1001/archneur.64.12.1721. PMID 18071034